CLINICAL TRIAL: NCT02830061
Title: An Interpretative Phenomenological Analysis Study Into the Experience of Teenagers and Young Adults Who Have Been Offered Ovarian Tissue Cryopreservation Prior to Cancer Treatment.
Brief Title: The Experience of TYAC Offered Ovarian Tissue Cryopreservation
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 12019
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Cancer; Fertility
Keywords: Cancer; Teenage; Young Adult; Fertility; Cryopreservation; Experience
MeSH Terms: conditions — Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TYAC: Teenagers and young adults who have received a cancer diagnosis which puts them at moderate-to-high risk of fertility impairment. Semi-structured interviews will take place with each individual participant.
  Interventions: Other: Interviews

INTERVENTIONS:
Other: Interviews — Individual semi-structured interviews for 30-60 minutes using an interview schedule developed from an interpretative phenomenological analysis framework.

SUMMARY:
This study looks at the experiences of teenagers and young adults who have been offered ovarian tissue cryopreservation prior to cancer treatment as a result of their cancer and/or cancer treatment putting them at moderate-to-high risk of premature ovarian failure.

DETAILED DESCRIPTION:
In the UK, around 2,200 teenagers and young adults (TYA) are diagnosed with cancer every year, and due to advances in treatments, survival rates have improved, with a current 5-year survival rate of more than 80%. This means there is a growing population of long-term survivors of childhood/adolescent cancer who may experience late effects of cancer and/or treatment. One such late effect is fertility impairment, which is a key issue for TYA with cancer. There are few clinical options currently available for the preservation of women's fertility in the UK; however, ovarian tissue cryopreservation (OTC) has been offered clinically at one primary treatment centre in the UK for the past 2-3 years. In an attempt to understand what it is like to be faced with potential infertility alongside a cancer diagnosis, previous studies have been conducted looking at young people's experiences of receiving, processing and living with this information, as well as their experiences of other FP techniques. However, no studies have looked at the experiences of cancer patients undergoing OTC. OTC differs to other FP options previously studied in several key ways, notably in that cancer treatment need not be delayed for it to go ahead, and it can be carried out with pre-pubertal females. This may mean that aspects of the process surrounding OTC are experienced differently to other FP options, and that OTC needs to be understood as a separate phenomenon. Although OTC is currently offered to women from birth to the age of 40 in the UK, the different experience of cancer and infertility across the lifespan necessitates a more specific focus for this study. TYA have been chosen as an understudied population, with more research needed to increase understanding of their unique psychosocial needs and their experience of health systems. Further, focusing on TYAC may capture individuals who have not started puberty and would therefore benefit from the introduction of this new technique by being unable to undergo other FP options.

The purpose of this research is therefore to take into account gaps in the literature and attempt to better understand the issues surrounding undergoing OTC for TYAC from the subjective experience of the individual.

ELIGIBILITY:
Inclusion Criteria:

* Aged 11-25 at time of procedure and aged 13+ at time of interview. Due to the short amount of time OTC has been available, there will be no time limit on how long ago the procedure took place.
* Received a cancer diagnosis carrying a moderate-high risk of premature ovarian failure as a result of the cancer and/or treatment.
* Have been offered ovarian cryopreservation by the ovarian cryopreservation service (participants will be included whether or not they have accepted the procedure).
* Has been confirmed as appropriate to approach by the consultant oncologist.

Exclusion Criteria:

* Under the age of 11 or over the age of 25 at time of procedure.
* Under the age of 13 at time of interview.
* Received a terminal diagnosis.
* The young person is unable to understand their diagnosis and/or fertility options, e.g. those with significant learning disabilities (guidance on this will be sought from the consultant oncologist as part of their approval).
* The young person is unaware that the procedure has taken place (guidance on this will be sought from the consultant oncologist as part of their approval).

Ages: 13 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: TYAC who have been offered OTC due to moderate-to-high risk of premature ovarian failure due to their cancer and/or cancer treatment.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Individual semi-structured interviews about the experiences of Teenagers and Young Adults with Cancer undergoing OTC | up to 60 min

CONTACTS AND LOCATIONS:
Overall Officials: Rebekah Tennyson, DClinPsy, Principal Investigator — Oxford Health NHS Foundation Trust